CLINICAL TRIAL: NCT00938951
Title: Evaluate the Ability of Systane Ultra to Improve Subjective Symptoms of Ocular Irritation Post 60 Min. Athletic Performance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SMA-09-22
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye Symptoms; Visual Performance
Keywords: Dry Eye; Visual Performance
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Systane® Ultra (Experimental): Systane® Ultra
  Interventions: Other: Systane® Ultra

INTERVENTIONS:
Other: Systane® Ultra — Polyethylene Glycol 400 0.4% / Propylene Glycol 0.3%

SUMMARY:
The primary objective of this study is to compare visual degradation in a stressed (forced stare) environment in patients before and after acute administration of Systane Ultra.

ELIGIBILITY:
Inclusion Criteria:

* Player/ Coach must answer "Yes" to the survey eligibility question.
* Player/Coach must voluntarily agree to participate in survey

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness of eye drop basd on athlete's opinion/experience during a one hour practice session | 60 minutes post-dosing with test article